CLINICAL TRIAL: NCT01035723
Title: Effect of Functional Genetic Polymorphisms on Brain Morphology
Brief Title: Effect of Functional Genetic Polymorphisms on Brain Morphology and Function
Status: Completed | Type: Observational
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999905406; 05-DA-N406
Record Dates: First submitted 2009-12-18; First posted 2009-12-21 (Estimated); Last update posted 2019-12-16 (Actual); Status verified 2013-02-25

CONDITIONS: Drug Abuse
Keywords: Prefrontal Cortex; Hippocampus; Amygdala; MRI; Cognitive Tasks
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Time Perspective: Other

SUMMARY:
Background:

- New research on genetics and the human genome has helped to identify certain genes that affect specific parts of the brain, including the parts that may be involved in drug use and dependency. Researchers are interested in studying both genetic information and brain activity to better understand variations in brain function among individuals.

Objectives:

- To study brain activity in conjunction with specific genetic information provided by healthy volunteers including smokers, non-smokers, people with drug dependence, and those who do not have any dependence on any substance.

Eligibility:

- Healthy volunteers between 18 and 50 years of age.

Design:

* This is an 8 10 hour study which may be completed in 1, 2, or 3 visits.
* Participants will complete questionnaires about emotional and psychological responses to different situations, including stressful situations.
* Participants will have a training session in a mock (fake) scanner to practice tasks to be completed in the real scanner.
* Participants will have the following two types of magnetic resonance imaging (MRI) scans in one scan session of the brain:
* A structural MRI scan to provide basic information about each participant's brain.
* A functional MRI scanning session, in which participants will perform a memory task to provide information about brain activity.
* Participants will provide blood samples for research and testing....

DETAILED DESCRIPTION:
Objective:

Functional genetic polymorphisms have been identified that influence the morphology and function of brain regions that have been implicated in addictive and neuropsychiatric disorders. This protocol aims to integrate genotyping with both structural and functional brain imaging to investigate the impact of specific functional polymorphisms on morphology and function of the amygdala and the hippocampus and on behavior mediated by these brain regions. Functional polymorphisms of the BDNF, SLC6A4, and DISC1 genes will be studied, as these are logical candidates to influence variability in brain morphology and function. The overall hypothesis is that variation in morphology and function of the amygdala and the hippocampus is explained, at least in part, by specific genotype differences.

Study Population:

The study population will consist of healthy male and female adult volunteers (18-50 years old).

Design:

After being medically cleared and giving written informed consent, each participant will undergo a structural MRI scan of the brain to be used for volumetric measurements of the amygdala, hippocampus, prefrontal cortex, and intracranial cavity. Each participant will undergo an fMRI scanning session, which will include an emotional context memory task specifically designed to require functioning of the amygdala and the hippocampus. A venous blood sample will be collected for genotyping of BDNF, SLC6A4, and DISC1 polymorphisms. Additionally, other functional polymorphisms that may influence brain structure may also be evaluated, in exploratory fashion. If participants have already had a blood sample collected for the genetics portion of another Neuroimaging Research Branch study, they may not need to have another sample taken.

Outcome Measures:

This protocol will provide no direct benefits to research participants. Understanding the relationship between genetic polymorphisms and brain morphology and their association to brain function and behavior may provide further clues to the neurobiological mechanisms underlying addictive and neuropsychiatric disorders. The potential risks are related to acquiring MRI scans in general. Medical supervision will be provided throughout the study.

ELIGIBILITY:
* INCLUSION CRITERIA:

To be eligible for this study, subjects must:

1. Be between the ages of 18 and 50.
2. Be in good health.
3. Be right handed.
4. Individuals with a substance abuse disorder may be included.

EXCLUSION CRITERIA:

Subjects will be excluded if they:

1. Are not suitable to undergo an MRI experiment due to pregnancy, implanted metallic devices (cardiac pacemaker or neurostimulator, some artificial joints, metal pins, surgical clips, or other implanted metal parts), body morphology, or claustrophobia.
2. Have coagulopathies, history of or current superficial or deep vein thrombosis, musculoskeletal abnormalities restricting an individual s ability to lie flat for an extended period of time.
3. Have HIV or syphilis.
4. Have a neurological illness to include, but not limited to, seizure disorders, migraine, multiple sclerosis, movement disorders, or history of head trauma, CVA, CNS tumor.
5. Have any current AXIS I psychiatric disorders including Attention Deficit Disorder (ADD). Have regular use of any prescription, over-the-counter, or herbal medication that may alter CNS function, cardiovascular function or neuronal-vascular coupling.
6. Have current dependence on any substance other than cocaine, marijuana, or nicotine.
7. Are cognitively impaired or are learning disabled.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 221 (Actual)
Dates: Start 2005-09-13; Study Completion 2013-02-25

PRIMARY OUTCOMES:
To understand the relationship between genetic polymorphisms and brain morphology and their association to brain function and behavior.

CONTACTS AND LOCATIONS:
Overall Officials: Elliot Stein, Ph.D., Principal Investigator — National Institute on Drug Abuse (NIDA)
Locations (1):
- National Institute on Drug Abuse, Baltimore, Maryland, United States

REFERENCES:
- [Background] Austin CP, Ma L, Ky B, Morris JA, Shughrue PJ. DISC1 (Disrupted in Schizophrenia-1) is expressed in limbic regions of the primate brain. Neuroreport. 2003 May 23;14(7):951-4. doi: 10.1097/01.wnr.0000074342.81633.63. PMID 12802181
- [Background] Bartzokis G, Altshuler LL, Greider T, Curran J, Keen B, Dixon WJ. Reliability of medial temporal lobe volume measurements using reformatted 3D images. Psychiatry Res. 1998 Apr 10;82(1):11-24. doi: 10.1016/s0925-4927(98)00007-9. PMID 9645547
- [Background] Bernstein DP, Stein JA, Newcomb MD, Walker E, Pogge D, Ahluvalia T, Stokes J, Handelsman L, Medrano M, Desmond D, Zule W. Development and validation of a brief screening version of the Childhood Trauma Questionnaire. Child Abuse Negl. 2003 Feb;27(2):169-90. doi: 10.1016/s0145-2134(02)00541-0. PMID 12615092